CLINICAL TRIAL: NCT03144024
Title: Comparison of Rigid Annuloplasty Ring With a Band in the Correction of Secondary Tricuspid Insufficiency
Acronym: BvsRR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BvsRR
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2016-09

CONDITIONS: Tricuspid Regurgitation
Keywords: Tricuspid Regurgitation; Insufficiency, Tricuspid Valve; Valvular Annuloplasty; Cardiac Valve Annulus Repair
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- band (Experimental)
  Interventions: Device: band implantation
- Rigid ring (Active Comparator)
  Interventions: Device: rigid ring implantation

INTERVENTIONS:
Device: band implantation
  Arms: band
Device: rigid ring implantation
  Arms: Rigid ring

SUMMARY:
randomized study which include comparison rigid ring and band devices in treatment tricuspid regurgitation.

DETAILED DESCRIPTION:
study include 308 patients. Patient will be randomized and 154 patient will receive band for treatment tricuspid regurgitation, rest patient will receive rigid ring. Follow up will be 1 year. Primary outcome - freedom of moderate or severe regurgitation. Secondary outcome - RV function, quality of life.

ELIGIBILITY:
Inclusion Criteria:

* moderate or severe tricuspid regurgitation

Exclusion Criteria:

* refusal to participate in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2016-09-14 (Actual); Primary Completion 2017-09-14 (Actual); Study Completion 2019-09-14 (Actual)

PRIMARY OUTCOMES:
tricuspid regurgitation | 12 months
death | 12 months

SECONDARY OUTCOMES:
right ventricle function | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- MeshalkinRI, Novosibirsk, Russia